CLINICAL TRIAL: NCT00694486
Title: Eustachian Tube Testing in a Pressure Chamber -- Validation
Brief Title: Eustachian Tube Testing in a Pressure Chamber -- Validation Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO07070157; 1P50DC007667 (NIH)
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2010-09

CONDITIONS: Otitis
Keywords: otitis; Eustachian tube function; Normal middle ear status
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy adult volunteers

SUMMARY:
This study will compare Eustachian tube function (ETF) testing in adults with intact tympanic membranes (TM) using a pressure chamber to that obtained using standard methods requiring a non-intact TM.

DETAILED DESCRIPTION:
The investigators propose to introduce new test methods and protocols to our laboratory for better clinical characterization of Eustachian tube function in ears with intact TM's. These test will be done in a pressure-chamber and will use previously published and newly developed methods. Participation will require a minimum of 5 visits to the ENT Research Center, 1 for myringotomy (putting a small hole in the eardrum) and 4 for ETF testing. Hearing testing will be done at entry and exit; otoscopy (looking at the ears) and tympanometry (a test done with an earplug and varying pressures in the ear canal) are done at every visit.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Normal middle-ear status

Exclusion Criteria:

* Chronic illness including asthma, pulmonary, or cardiac problems
* Pregnancy
* >10 dB hearing loss in any of the speech frequencies
* Past history of sensitivity or allergic reaction to lidocaine or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Eustachian tube function testing results | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William J Doyle, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- ENT Research Center Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States